CLINICAL TRIAL: NCT03408769
Title: Metastatic Breast Carcinoma: Evaluation of Women Sexual Quality of Life
Brief Title: Metastatic Breast Carcinoma and Women Sexual Quality of Life
Acronym: SexoMBC
Status: Completed | Type: Observational
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A03413-50
Record Dates: First submitted 2018-01-18; First posted 2018-01-24 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Metastatic Breast Carcinoma
Keywords: Cancer; Sexuality; Quality of life; Intimacy; BISF-WBrief Index of Sexual Functioning for Women questionnaire; Quality of life questionnaire (EORTC QLQ-BR23):; Partnership questionnaire (partnerschaftsfragebogen; PFB)
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Sexuality; pseudofolliculitis barbae

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Medical questionnaire — * Brief Index of Sexual Functioning for Women questionnaire
  * Quality of life questionnaire (EORTC QLQ-BR23)
  * Partnership questionnaire (partnerschaftsfragebogen; PFB)
  * Short interview about their sexual intimacy

SUMMARY:
Sexual health is one of the relevant parameters for assesing the quality of life.

Improvement sexual and emotional function improves quality of life scores and depression or anxiety in curative phase.

The purpose of the study is to assess the quality of sexual life of postmenopausal women with metastatic breast cancer in couples and to establish links with overall quality of life and the quality of the relationship.

DETAILED DESCRIPTION:
We use a quantitative methodology to assess quality of female sexual life, quality of life and quality o relationship with validated scientific questionnaires.

The sexual and emotional intimacy will be explored by semi structured interview, not mandatory for patients.

ELIGIBILITY:
Inclusion Criteria:

* Women with metastatic breast cancer
* Age ≥ 50 and < 70 years old
* Diagnosis of metastatic breast cancer at least 6 months prior to study participation
* Patient living with a partner
* Menopausal women (absence of menstruation for 1 year minimum)
* ECOG performance status ≤ 2
* Affiliated to public health system
* Informed and having expressed her non-opposition

Exclusion Criteria:

* Patient in exclusive palliative care
* Single or not living in a couple
* Non-menopausal patient

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be offered to women aged 50 to 70, with metastatic breast carcinoma and living in a couple and followed at the Lorraine Institute of Oncology.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-04-04 (Actual)

PRIMARY OUTCOMES:
Quality of sexual life of postmenopausal women with metastatic breast carcinoma living in couples | 1 day
  Quality of sexual life will assessed by BISF-W (Brief index of sexual functioning for women) questionnaire

SECONDARY OUTCOMES:
Quality of life | 1 day
  Quality of life will assessed by quality of life breast cancer module questionnaire (QLQ-BR23) (Hinz et al, 2014)
Quality of Relationship of the couple | 1 day
  Quality of Relationship of the couple will assessed by partnership questionnaire (PFB). 30 items making up a global scale measuring the Quality of relationship (PFB).Quality of relationship (PFB) score can be obtained with the following equation: PFB = (30 - Quarreling) + Tenderness + Togetherness/communication ( Rossier et al, 2006).
Sexual and emotional intimacy | 1 day
  Patients will be interviewed by open-ended questions face to face concerning their Sexual and emotional intimacy.

CONTACTS AND LOCATIONS:
Overall Officials: Dubuc Myriam, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, France